CLINICAL TRIAL: NCT00005869
Title: Phase III Randomized Study of RFS 2000 (9-Nitro-Camptothecin, 9-NC) Versus Gemcitabine HCl in Chemonaive Pancreatic Cancer Patients
Brief Title: Nitrocamptothecin Compared With Gemcitabine in Treating Patients With Unresectable Locally Advanced or Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067905; SUPERGEN-RFS2000-02
Record Dates: First submitted 2000-06-02; First posted 2004-02-25 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2007-06

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; rubitecan

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: rubitecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether nitrocamptothecin is more effective than gemcitabine for pancreatic cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of nitrocamptothecin with gemcitabine in treating patients who have unresectable locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall survival, time to treatment failure, clinical benefit response rate (analgesic consumption, pain intensity, performance status, and weight change), and objective response rate in chemotherapy-naive patients with unresectable locally advanced or metastatic adenocarcinoma of the pancreas treated with oral nitrocamptothecin vs gemcitabine. II. Compare the toxicity of these 2 regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to measurable disease (yes vs no), Karnofsky performance status (50-70% vs 70-100%), and prior radiotherapy. Patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive oral nitrocamptothecin on days 1-5. Treatment repeats every week for 8 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease after week 8 may receive additional courses. Arm II: Patients receive gemcitabine IV over 30 minutes on day 1. Treatment repeats every week for 7 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo 1 week of rest. Patients with stable or responding disease after week 8 may receive gemcitabine IV over 30 minutes on days 1, 8, and 15. Courses repeat every 4 weeks. Pain is assessed within 7 days prior to study, at days 28 and 56 during study, and then every 28 days after completion of study. Patients are followed every 3 months for 1 year or until death.

PROJECTED ACCRUAL: Approximately 994 patients (497 per arm) will be accrued for this study within 22 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed unresectable locally advanced (stage II or III) or metastatic (stage IV) adenocarcinoma of the pancreas

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: Granulocyte count greater than 1,500/mm3 Hemoglobin at least 9 g/dL Platelet count greater than 100,000/mm3 Hepatic: SGOT and SGPT no greater than 3 times normal (5 times normal if liver tumor present) Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior immunotherapy and recovered No filgrastim (G-CSF) concurrent with nitrocamptothecin Concurrent epoetin alfa allowed Chemotherapy: Prior fluorouracil as radiosensitizer allowed No other prior chemotherapy (e.g., nitrocamptothecin or gemcitabine) No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal or corticosteroid therapy Patients requiring hormonal therapy or corticosteroid therapy for medical reasons may remain on study, but will not be evaluable for clinical benefit response Radiotherapy: At least 3 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: See Disease Characteristics More than 2 weeks since prior major surgery and recovered Prior stent placement allowed No planned surgery within 8 weeks after initiation of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-11

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A. Romel, MS, Study Chair — Astex Pharmaceuticals, Inc.
Locations (1):
- SuperGen, Incorporated, Dublin, California, United States